CLINICAL TRIAL: NCT06200155
Title: TRIP - TReatment to Improve Depression and/or Anxiety Using Psilocybin-Assisted Psychotherapy in Patients With Advanced Cancer on Maintenance Therapy
Brief Title: Psilocybin-Assisted Psychotherapy in Patients With Advanced Cancer on Maintenance Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2022-0170; NCI-2023-11090 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Depression, Anxiety; Psilocybin-Assisted Psychotherapy; Advanced Cancer
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Psilocybin; Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Participants will receive psilocybin (25 mg).
  Interventions: Drug: Psilocybin
- Arm B (Placebo Comparator): Participants will receive the placebo (100 mg of Niacin).
  Interventions: Other: Niacin

INTERVENTIONS:
Drug: Psilocybin — Given by PO
  Arms: Arm A
Other: Niacin — Given by PO
  Arms: Arm B

SUMMARY:
To learn about the feasibility, safety, and effects of psilocybin-assisted psychotherapy on depression and/or anxiety in participants who are being treated for advanced cancer.

DETAILED DESCRIPTION:
Primary Objective

To examine the feasibility, safety, effect size estimates of psilocybin-assisted psychotherapy for participants with depression and/or anxiety who are being actively treated for advanced cancer. Feasibility will be measured as: At least 20% of eligible participants consent and at least 60% of consented participants complete the two doses of treatment.

Secondary Objectives

1. Determine whether psilocybin-assisted psychotherapy improves measures of quality of life (e.g., sleep, pain, functional status) and psychosocial well-being (e.g., finding meaning and post-traumatic growth), as measured by the following: PHQ-9, GAD-7, PROMIS-10, PROMIS-A, PROMIS-D, MEQ30 (mystical experience), Flourishing scale, mDES, 5D-ASC (altered states), and Posttraumatic Growth Inventory.
2. Determine whether psilocybin-assisted psychotherapy improves functional status per clinician-rated outcome measures.
3. Assess the effects of psilocybin-assisted psychotherapy on cancer treatment adherence determined by the likelihood that participants will follow the prescribed treatment (adherence) and continue the treatment for the duration prescribed (persistence) for these maintenance therapies.
4. Measure the change in inflammatory markers (IL6, TNF, and CRP) and in frequency and activation status of peripheral immune cell populations assessed by immune monitoring through flow cytometry.
5. Examine changes in central nervous system plasticity through the use of fMRI, specifically changes in 5-HT2A-rich and higher-order functional networks, as well as a global increase in brain network integration.
6. Evaluate the Impact on MDASI measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have one of the following histology documented tumor types: non-small cell lung carcinoma, renal cell carcinoma, urothelial carcinoma, prostate cancer, head and neck squamous cell carcinoma, ovarian cancer, breast cancer, gastric/GEJ cancer, cervical, anal, or MSI-high
2. Documentation of locally advanced, recurrent, or metastatic incurable malignancy that has partially responded or progressed after at least 1 available standard therapy and disease is stable (no progression of disease for 3 months or more on current treatment regimen)
3. No prior grade 3 AEs on current standard of care cancer treatment regimen;
4. Age ≥ 25 years; as by the age of 25 brain is fully developed.
5. Have a DSM-V psychiatric diagnosis, as determined by the SCID (Structured Clinical Interview for DSM, by a board certified psychiatrist), of one or more of the following Axis I psychiatric disorders that is judged to have been precipitated by the psychological stress of the cancer diagnosis: Generalized Anxiety Disorder; Acute Stress Disorder; Posttraumatic Stress Disorder; Major Depressive Disorder; Dysthymic Disorder; Adjustment Disorder with Anxiety; Adjustment Disorder with Depressed Mood; Adjustment Disorder with Mixed Anxiety and Depressed Mood; Adjustment Disorder with Disturbance of Conduct; Adjustment Disorder with Disturbance of Emotions and Conduct. Psychiatric diagnosis are determined by a MD Anderson board certified psychiatrist.
6. At least 6 months life expectancy as per primary medical oncologist.
7. Have an ECOG performance status of 0, 1, or 2.
8. Must have no major cognitive impairment and be oriented to person, place, and time (e.g. mini mental exam).
9. Must demonstrate willingness to travel to MD Anderson Cancer center for all treatment and follow-up sessions, as well as consent to complete all evaluation instruments and assessments.
10. Agree to abstain from any nicotine products for at least 12 hours prior to psilocybin administration until approximately 12 hours after (or when all post-session questionnaires have been completed) as well as on days of salivary sample collection.
11. Refrain from any psychoactive drugs (including alcohol) for 48 hours prior to psilocybin sessions (except as described above for nicotine and caffeine) and must refrain from psychoactive drugs 12 hours after psilocybin sessions. Must consent to urine drug screen (UDS) which will be given before receiving psilocybin. Participants with positive drug test will be retested (UDS) after 6 weeks and included if the repeated UDS is negative. Participant tested positive for a prescribed substance are eligible. Participant failing on the 2nd test (UDS) will be excluded.
12. Must be free from any regularly scheduled psychotropic (antidepressant/anxiolytic class) medications and those with primary MOA on serotonergic neurons (e.g., ondansetron) for a minimum of 2 weeks prior to study or 4 weeks for SSRI. Intermittent or PRN use of short-acting anxiolytics may be permitted as defined below in exclusionary criteria).
13. Inhibitors of monoamine oxidase, UGT1A9, 1A10, and aldehyde or alcohol dehydrogenase should be discontinued 5 half-lives prior to active dose of psilocybin.
14. Eligible participants will have a responsible individual that will provide transportation home after the psilocybin session is complete.
15. Fluent in English

Exclusion Criteria:

1. History of depression prior to cancer diagnosis.
2. Clinically significant suicidality or high risk of completed suicide defined as:

   i. Answer 'Yes' to C-SSRS Suicidal Ideation items 4 or 5 within the last 2 months at Screening or 'since last visit' at Baseline ii. Report having had any C-SSRS Suicidal Behavior item within the past 12 months at Screening or 'since last visit' at Baseline, as defined by 'Yes' to any of the following on the C-SSRS: actual attempt, interrupted attempt, aborted attempt, or preparatory acts iii. Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of suicidal or self-injurious behavior
3. History of bipolar disorder, psychosis (of any nature), and seizures.
4. Functionally limiting comorbid conditions such as second primary malignancies in CNS or chest, and history of total laryngectomy or total .glossectomy.
5. ECG with QTc > 450.
6. Patients with metal implants.
7. Asymptomatic ALT or AST elevations >/= 5X upper limit of normal, symptomatic ALT or AST elevations >/= 2X upper limit of normal, or total bilirubin >/= 2X upper limit of normal.
8. The effects of psilocybin on the developing human fetus are unknown. For this reason, pregnant women will be excluded (Urine test for screening), women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the participant presents with an applicable exclusionary factor which may be one of the following:

   Postmenopausal (no menses in greater than or equal to 12 consecutive months). History of hysterectomy or bilateral salpingo-oophorectomy. Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).

   History of bilateral tubal ligation or another surgical sterilization procedure.

   Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
9. persons with first- or second-degree relatives who have schizophrenia or other psychotic disorders, or bipolar I or II disorder.
10. Actively progressing disease as defined by the primary oncologist.
11. Vulnerable populations, including children and cognitively impaired patients, will not be enrolled in this study.
12. Participants with brain metastases.
13. Risk for hypertensive crisis defined as Screening, Baseline, and Medication Session (prior to dosing) Blood Pressure >140/90 mmHg and HR> 90 bpm.
14. Unstable medical conditions or serious abnormalities of complete blood count, chemistries, or ECG that in the opinion of the study physician would preclude safe participation in the trial. Some examples include:

    i. Uncompensated congestive heart failure ii. Clinically significant arrhythmias (e.g., ventricular fibrillation, torsades) or clinically significant ECG abnormality (i.e., QTC interval > 450) iii. Recent acute myocardial infarction or evidence of ischemia iv. Malignant hypertension v. Congenital long QT syndrome vi. Acute renal failure vii. Severe hepatic impairment viii. Respiratory failure
15. Significant central nervous system (CNS) pathology. Some examples include:

    i. Primary or secondary cerebral neoplasm ii. Epilepsy iii. History of stroke iv. Cerebral aneurysm v. Dementia vi. Delirium
16. a. High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation. Examples include: i. Agitation ii. Violent behavior b. Active substance use disorders (SUDs) defined as: DSM-5 criteria for moderate or severe alcohol or drug use disorder (excluding caffeine and nicotine) within the past year c. Extensive use of serotonergic hallucinogens (e.g., LSD, psilocybin) defined as: i. Any use in the last 12 months ii. >25 lifetime uses d. History of hallucinogen persisting perception disorder (HPPD) e. Concurrent Medications i. Antidepressants ii. Centrally-acting serotonergic agents (e.g., MAO inhibitors) iii. Antipsychotics (e.g., first and second generation) iv. Mood stabilizers (e.g., lithium, valproic acid) v. Aldehyde dehydrogenase inhibitors (e.g., disulfiram) vi. Significant inhibitors of UGT 1A0 or UGT 1A10 vii. Niacin. Note: If taking any supplement containing niacin, agrees to suspend use for at least five days prior to dosing and for the duration of the study f. Have a positive urine drug test including Amphetamines, Barbiturates, Buprenorphine, Benzodiazepines, Cocaine, Cannabis, Methamphetamine, MDMA, Methadone, Opiates (Morphine, Oxycodone), Phencyclidine (PCP), and Tetrahydrocannabinol (THC).

    i. Note: Prescribed opiate medications (e.g., cancer-related pain) will be allowed to continue through the study period for participants who have been on a stable dose of such medicine for at least 1 month prior to Screening, as determined during review of concomitant medications.

    ii. Note: Prescribed benzodiazepine medications and nonbenzodiazepine sleeping medications will be allowed to continue through the study period for participants who have been on a stable dose of such a medicine for at least 6 weeks prior to Screening, as determined during review of concomitant medications.

    iii. Note: Participants using cannabis, including legal cannabis, for any purposes must agree to refrain from use beginning at Screening, as confirmed with a negative Baseline drug test, and through to the end of the study.

    iv. Note: Participants using prescribed psychostimulants (amphetamines and Ritalin), must agree to refrain from use two weeks prior to baseline visit, as confirmed with a negative Baseline drug test, and through to the end of the study.

    g. Have a psychiatric condition judged to be incompatible with establishment of rapport with the study therapists or safe exposure to psilocybin h. Have any psychological or physical symptom, medication or other relevant finding prior to randomization, based on the clinical judgment of the PI or relevant clinical study staff that would make a participant unsuitable for the study.

    i. Have an allergy or intolerance to any of the materials contained in either drug product j. Be enrolled in another clinical trial assessing intervention(s) for anxiety, depression, and/or existential distress (e.g., pharmacologic or psychotherapeutic interventions)
17. Participants who have any of the below niacin contraindications:

    1. Active liver disease or unexplained persistent elevations in hepatic transaminases
    2. active peptic ulcer disease
    3. arterial bleeding
    4. Hypersensitivity to niacin or any component of this medication
18. BP> 200/110 (or malignant hypertension defined as 200/120) would prevent a patient from receiving psilocybin dosing and would prompt calling a physician during blood pressure monitoring for cardiac risk evaluation.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Moran Amit, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-12-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT06200155/ICF_000.pdf